CLINICAL TRIAL: NCT07392476
Title: Continuous Glucose Monitoring in Polycystic Ovarian Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 25-679
Record Dates: First submitted 2025-12-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Polycystic Ovarian Syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Polycystic Ovarian Syndrome: Patients with Polycystic Ovarian Syndrome
  Interventions: Device: Stelo glucose biosensor by Dexcom

INTERVENTIONS:
Device: Stelo glucose biosensor by Dexcom — Unblinded continuous glucose monitoring (CGM) system

SUMMARY:
The purpose of this study is to learn more about blood sugar control in polycystic ovarian syndrome.

The patient will be asked to wear a continuous glucose monitor (CGM) device that is applied to the arm with a sensor or filament that goes under the skin to measure your sugar levels. The patient will wear this at certain time points throughout the study. There will have a total of 2 blood draws (about 1 tsp. of blood) at screening and the 6-month visit, a measure of the patients body muscle and fat (body composition), and fill out a questionnaire at the end of the first 3 months and 6 months.

Study participation in the research will last about 6 months.

ELIGIBILITY:
Inclusion Criteria

1. Adult 18-45 years old
2. Diagnosis of PCOS by usual clinical method such as by Rotterdam criteria
3. BMI >25 kg/m2

Exclusion Criteria

1. Currently on medications that can improve glucose levels such as metformin and glucagon-like receptor 1 agonists (GLP1RA)
2. Previously intake of above-mentioned medications but less than 3 months since last intake of metformin or less than 6 months since last intake of GLP1RA
3. Currently on insulin
4. Does not have Stelo-compatible phone
5. Fasting glucose >100 mg/dL (because that is the cutoff for prediabetes) (either labs taken within a week after first visit or within 3 months before start of study
6. HbA1c > 5.7% (because this is the cutoff for prediabetes) (either labs taken after screening visit or within 3 months before start of study)
7. History of anorexia or bulimia
8. Current or previous CGM use
9. Use of oral contraceptives at time of enrolment
10. Intent to become pregnant within 6 months (will need to terminate study if gets pregnant as glucose readings will be affected)
11. Menopausal women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with polycystic ovarian syndrome (PCOS).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Continuous Glucose measure derived glucometrics | 6 months
  To describe CGM-derived glucometrics in patients with PCOS before and after lifestyle modification and/or pharmacologic intervention.
Continuous Glucose measure derived glucometrics and Polycystic ovarian syndrome | 6 months
  To explore associations between CGM-derived glucometrics and PCOS-related clinical markers such as anti-mullerian hormone (AMH), HbA1c, lipid levels, body mass index, and body composition. Associations between glucometrics and PCOS-related clinical markers will be evaluated using correlations, two-sample t-tests or Pearson chi-square tests, as appropriate.
Lifestyle behaviors | 6 months
  To evaluate patient perception of CGM in influencing lifestyle behaviors. The survey includes 5 multiple choice questions and will be summarized using frequencies and percentages.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No